CLINICAL TRIAL: NCT06201871
Title: Effect of Alcohol Consumption on the Success Rates of Local Anesthesia in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Effect of Alcohol Consumption on the Success Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IANB
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcoholic patients (Experimental): Patients will receive an inferior alveolar nerve block injection using 1.8 mL of 2% lidocaine with 1: 80 000 epinephrine using a direct Halsted approach.
  Interventions: Drug: Lidocaine Hydrochloride
- Control patients (Active Comparator): Patients will receive an inferior alveolar nerve block injection using 1.8 mL of 2% lidocaine with 1: 80 000 epinephrine using a direct Halsted approach.
  Interventions: Drug: Lidocaine Hydrochloride

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Patients will receive an inferior alveolar nerve block injection using 1.8 mL of 2% lidocaine with 1: 80 000 epinephrine using a direct Halsted approach.

SUMMARY:
This prospective, randomized, double-blind clinical trial will be carried out Conservative Dentistry, Faculty of Dentistry, Jamia Millia Islamia. Seventy adult patients (35 alcoholic and 35 non-alcoholics) with symptomatic irreversible pulpits in a mandibular first or second molar will receive an IANB with 2% lidocaine. In case of pain during treatment, the procedure will be stopped, and the patients will be asked to rate the pain on the Heft-Parker scale. The injection shall be considered as successful if the patient reports pain scores less than 55 on the HP scale.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic carious exposed mandibular first or second molars.
* Alcoholic patients: Patient with low-moderate drinking levels according to the US National Institute on Alcohol Abuse and Alcoholism
* Control patients: No history of alcohol consumption
* Positive and prolonged response to thermal sensitivity tests and electric pulp test.
* Vital coronal pulp on access cavity preparation.
* American Society of Anesthesiologists class I or II medical history.
* Ability to understand the use of pain scales.

Exclusion Criteria:

* Active pain in more than 1 teeth
* Teeth with fused roots.
* Radiographic evidence of an extra root.
* Large restorations with overhanging margins.
* Full crowns or deep periodontal pockets.
* Hypertension or cardiovascular diseases, compromised immunity, active infection or inflammation
* Known allergy or contraindications to any content of the local anesthetic solution or non-steroidal anti-inflammatory drugs (NSAIDs)
* History of known or suspected drug abuse.
* Taking any drugs which could affect the pain perception, e.g, opioids, antidepressants, anticonvulsants, muscle relaxants, anxiolytics, sedatives, nsaids. 23
* Pregnant or breastfeeding patients.
* Patients with asthma, gastric ulcers, bleeding disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
Anesthetic success | 15 minutes following the injection
  The injection shall be considered as successful if the patient reports pain scores less than 55 on the visual analouge scale. The scale is 170mm long, with 0 marked as no pain and 170 marked as the maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Jamia MIliia Islamia, New Delhi, India

IPD SHARING:
Plan to Share IPD: No